CLINICAL TRIAL: NCT05486013
Title: A Prospective, Open, Multicenter Clinical Observational Study of Zanubrutinib in the Treatment of Recurrent Refractory Mantle Cell Lymphoma
Brief Title: Zanubrutinib in the Treatment of Recurrent Refractory Mantle Cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Peking Union Medical College Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other); China-Japan Friendship Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022276
Record Dates: First submitted 2022-07-04; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-06

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
80% of patients with mantle cell lymphoma (mantle cell lymphoma, MCL)were in the advanced tumor stage when they were first diagnosed. Zabutinib, as a new generation of BTK inhibitors, has better targeting and safety in clinical application. Previous studies have confirmed that zabutinib has good efficacy in treating relapsed refractory MCL. However, for patients with a high risk of drug resistance to BTK inhibitors or patients with drug resistance, the efficacy of BTK inhibitors alone is poor, and combined therapy can improve the poor prognosis of these patients. Therefore, the primary purpose of this study is to evaluate the safety and efficacy of zebutenil in treating recurrent, refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
Mantle cell lymphoma (mantle cell lymphoma, MCL) is a kind of B-cell lymphoma with unique histomorphology, immunophenotype, and cytogenetic characteristics, accounting for 6% of non-Hodgkin's lymphoma. It usually occurs in older adults, with a median age of 68. In recent years, although the application of new drugs has made much progress in the treatment of mantle cell lymphoma, the overall curative effect is not good. The vast majority of patients relapse after treatment. The median survival time is 3-5 years due to a lack of standard treatment. MCL responds to combined therapy, but easy recurrence is still problematic in clinical treatment. 50% to 60% of MCL eventually relapsed after treatment. Among them, BTK inhibitors exert their anti-tumor activity by promoting apoptosis and inhibiting tumor cell proliferation, inhibiting chemokine from blocking B cell migration, and reducing tumor B cell adhesion, which has become a milestone in the treatment of recurrent, refractory MCL. Zabutinib, as a second-generation BTK inhibitor, optimizes its chemical structure. Compared with the first-generation BTK inhibitor, zabutinib has complete and lasting BTK inhibition, more accurate targeting selection, and better clinical application safety. Previous clinical studies have shown that BTK inhibitor zabutinib is effective in treating recurrent and refractory MCL. However, using BTK inhibitors alone to produce drug resistance will cause rapid tumor growth in MCL patients, which has always been a difficulty in clinical treatment. A retrospective analysis of 693 Chinese patients with MCL showed that the complete remission rate (CR） of the initial treatment of MCL in China was 40.9%, the objective remission rate（ORR） was 81.6%, the 5-year progression-free survival rate(PFS) was 51.2%, and the 5-year overall survival time (OS) was 58.4%. It is significantly lower than the curative effect on foreign patients. At the same time, 56.8% of the patients relapsed after remission, so the treatment plan for patients in the Chinese population needs to be further optimized. Currently, the clinical application of zabutinib combined with ortozumab, a BCL-2 inhibitor, dexamethasone, and pomalidomide is one of the therapeutic regimens for recurrent refractory MCL with a high complete remission rate and safety. In order to better collect the clinical data on zabutinib combination therapy and make a more scientific and accurate evaluation, this study carried out a clinical observation study on the safety and efficacy of zabutinib combination therapy in recurrent refractory MCL. The survival index was evaluated by the objective remission rate (ORR) of 2 and 4 cycles of the combination regimen, and the adverse reactions and recurrence rates were collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been enrolled in other clinical trials.
2. Patients who are receiving immunosuppressive therapy for other diseases.
3. Patients who have received other treatments for lymphoma before joining the group.
4. Complicated with other malignant tumors.
5. The researchers determined that the patients were not suitable for the study.
6. Severe mental or neurological disorders that affect informed consent or expression of adverse reactions.
7. Patients who cannot be followed up.

Exclusion Criteria:

1. Patients who have been enrolled in other clinical trials.
2. Patients who are receiving immunosuppressive therapy for other diseases.
3. Patients who have received other treatments for lymphoma before joining the group.
4. Complicated with other malignant tumors.
5. The researchers determined that the patients were not suitable for the study.
6. Severe mental or neurological disorders that affect informed consent or expression of adverse reactions.
7. Patients who cannot be followed up.

Exit (drop-off) criteria :

1. Subject requires to quit.
2. Serious adverse events occurred during the trial, so it is inappropriate to continue the trial.
3. Due to the progression of the disease during the trial, it is not appropriate to continue to use the trial drugs and / or to continue this study program.
4. Incomplete research data records.
5. Patients who cannot be followed up.

Withdrawal cases should be retained for future reference and transferred from the last record to the final record for ITT analysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with recurrent refractory mantle cell lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-05-26 (Estimated); Study Completion 2025-11-26 (Estimated)

PRIMARY OUTCOMES:
The objective response rate | From the time of the first drug administration until the end of two cycles (each cycle is 28 days)
  This trial's primary outcome is the objective response rate (ORR) of two cycles of treatment

SECONDARY OUTCOMES:
The negative rate of minimal residual disease | From the first day of medication to the end of 1 year
  The secondary outcome of this trial is 1-year negative rate of minimal residual disease(MRD)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China